CLINICAL TRIAL: NCT05737992
Title: The Effect of of High Intensity Interval Training in Water on Functional Fitness in People With Parkinson's Disease: A Randomized Controlled Trial
Brief Title: The Effect of Exercise in Water on Functional Fitness in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pardis Specialized Wellness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PA21PD-2-02
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Parkinson; Parkinson Disease; Neurologic Disorder
Keywords: Parkinson Disease; Aqua Therapy; Balance; Neurological Disorders
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases | interventions — Exercise; Water

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocate to intervention group or control group and will be examined in the same way
Who Masked: Outcomes Assessor
Masking Description: A research project collaborator who is not informed about grouping of participants will obtain outcome measurements of the functional tests. Outcome adjudicators and data analysts will be kept blinded to the allocation. Moreover, all investigators, staff, and participants will be kept masked to outcome measurements and trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients in the intervention group will do high intensity interval training (HIIT) in water. In this study, HIIT training will be short intervals (30 seconds) of movements and 15 seconds of rest.Exercises will be done in a floating position in the deep part. The intervention will be done 3 sessions weekly. The length will be 8 weeks.
  Interventions: Other: Exercise in water
- Control group (No Intervention): The patients will continue their usual medication and their usual physical activity.

INTERVENTIONS:
Other: Exercise in water — Participants will do some exercises in water for 30-60 minutes. Exercises will be performed at a moderate exercise intensity (12-14 on the Borg Rate of Perceived (RPE) Scale).
  All protocols are tailor-made based on each individual's needs and physical abilities.
  Arms: Exercise group

SUMMARY:
The goal of this clinical trial study is to learn about the effect of aquatic exercise in parkinson's patients. The main questions it aims to answer are:

* What is the effect of exercise in water on balance in parkinson's patients?
* What is the effect of exercise in water on muscle strength in parkinson's patients?
* What is the effect of exercise in water on flexibility in parkinson's patients? Parkinson's patients in this study will do some functional tests. One group of them will do exercises in water 3 times weekly for 8 weeks.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive, neurodegenerative movement disorder characterised by the motor symptoms bradykinesia, tremor, rigidity, and postural instability. These are commonly associated with non-motor disturbances, neurobehavioural symptoms and reduced quality of life.

Exercise is currently recommended as an additional strategy to manage PD-induced disability and is a key component of rehabilitation programs for people with PD.

Aquatic exercise is another form of non-conventional exercise that has been growing in popularity in the context of neurorehabilitation.16 The aquatic setting offers specific mechanical advantages due to the hydrostatic and hydrodynamic principles of buoyancy, viscosity and drag.

Due to its ability to enhance functional mobility whilst also being enjoyable,aquatic exercise has become a very popular form of physical training in the management of neurodegenerative disorders.

Recent studies suggest that high-intensity interval training (HIIT) is promising for promoting neuroplasticity in human PD, with short training time and reduced burden. Biomarkers for neuroplasticity such as brain-derived neurotrophic factor (BDNF) and neurodegeneration (including neurofilament light chain ((NfL) and α-synuclein) may play a role, but their response to HIIT is not well-investigated.

The aims of this study are to investigate the effects of HIIT exercises in water on balance, muscle strength, flexibility and gait speed in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of idiopathic PD, from mild to moderate stages (severity from 1 to 4), according to the original version of the Hoehn & Yahr scale (HY)17, assessed by the neurologist
* Having medical certificate for performing physical activities and attending heated pools

Exclusion Criteria:

* Having another neurological pathology
* Having limiting orthopedic or heart associated conditions
* changing physical activities or L-dopa-based drug intake parameters

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Rate of changes of Balance | Pre test and posttest (after 8 weeks)
  Balance will be assessed by Berg Balance Scale test
Rate of changes of Flexibility | Pre test and posttest (after 8 weeks)
  Balance will be assessed by Sit & Reach test
Rate of changes of Muscle Strength | Pre test and posttest (after 8 weeks)
  Balance will be assessed by 30 s Sit to Stand test and Arm Curl test
Rate of changes of Gait Speed | Pre test and posttest (after 8 weeks)
  Balance will be assessed by 4-meters gait speed test

CONTACTS AND LOCATIONS:
Overall Officials: MohammadAli Tabibi, Study Director — Head of Department
Locations (1):
- Pardis specialized wellness institute, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification are to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the paper is published. No end date.
Access Criteria: Data will be accessible with no criteria. Anyone who wishes will have access to data.

REFERENCES:
- [Result] Methajarunon P, Eitivipart C, Diver CJ, Foongchomcheay A. Systematic review of published studies on aquatic exercise for balance in patients with multiple sclerosis, Parkinson's disease, and hemiplegia. Hong Kong Physiother J. 2016 Jul 7;35:12-20. doi: 10.1016/j.hkpj.2016.03.002. eCollection 2016 Dec. PMID 30931029
- [Result] Hughes AJ, Daniel SE, Lees AJ. Improved accuracy of clinical diagnosis of Lewy body Parkinson's disease. Neurology. 2001 Oct 23;57(8):1497-9. doi: 10.1212/wnl.57.8.1497. PMID 11673599
- [Result] Cugusi L, Cadeddu C, Nocco S, Orru F, Bandino S, Deidda M, Caria A, Bassareo PP, Piras A, Cabras S, Mercuro G. Effects of an aquatic-based exercise program to improve cardiometabolic profile, quality of life, and physical activity levels in men with type 2 diabetes mellitus. PM R. 2015 Feb;7(2):141-8; quiz 148. doi: 10.1016/j.pmrj.2014.09.004. Epub 2014 Sep 10. PMID 25217820
- [Result] Jimenez-Maldonado A, Renteria I, Garcia-Suarez PC, Moncada-Jimenez J, Freire-Royes LF. The Impact of High-Intensity Interval Training on Brain Derived Neurotrophic Factor in Brain: A Mini-Review. Front Neurosci. 2018 Nov 14;12:839. doi: 10.3389/fnins.2018.00839. eCollection 2018. PMID 30487731
- [Result] Hirsch MA, van Wegen EEH, Newman MA, Heyn PC. Exercise-induced increase in brain-derived neurotrophic factor in human Parkinson's disease: a systematic review and meta-analysis. Transl Neurodegener. 2018 Mar 20;7:7. doi: 10.1186/s40035-018-0112-1. eCollection 2018. PMID 29568518